CLINICAL TRIAL: NCT05560321
Title: Measuring the Impact of an Enhanced Strategy for Daily Disinfection in Acute Care Hospital Rooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: PDI Healthcare Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro00103576
Record Dates: First submitted 2022-09-22; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Disinfection
Keywords: Disinfection, contamination

STUDY DESIGN:
Intervention Model Description: Each participant's inpatient room was enrolled in both the intervention and control arms at the same time.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind - exception of the study team member applying the disinfectant product (intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Application of a 24-hour continuously acting quaternary ammonium salt disinfectant: Sani24 (PDI Healthcare Inc.) by study team
  Interventions: Other: Sani24; Other: Routine Disinfection
- Control (Active Comparator): Routine disinfection completed by hospital staff
  Interventions: Other: Routine Disinfection

INTERVENTIONS:
Other: Sani24 — Disinfectant
  Arms: Intervention
Other: Routine Disinfection — Routine disinfection at the study hospital

SUMMARY:
To determine the effectiveness of an enhanced strategy for daily disinfection in acute care hospital rooms comparing the addition of sani24 to routine daily cleaning versus the control of routine daily cleaning.

DETAILED DESCRIPTION:
The study Investigator will evaluate the effectiveness of a) adding sani24 to the standard daily cleaning and b) routine daily disinfection in acute care hospital rooms to measure the reduction in bioburden. In other words, the study aims to answer the following research question: does the addition of an additional disinfection technology (Sani24) decrease the environmental bioburden in inpatient hospital compared to routine disinfection?

This trial was conducted in acute care hospital rooms at Duke University Hospital in Durham, North Carolina from November 2021 to March 2022. Room surfaces were divided in two (e.g., right vs. left), allowing each patient room to serve as its own control. The intervention was a quaternary ammonium salt-based 24-hour continuously active germicidal wipe, Sani-24 (PDI Healthcare, Woodcliff, NJ) that was applied in addition to routine disinfection. The control arm received no intervention beyond routine disinfection. Environmental services were blinded to study arms and no changes to routine cleaning protocols occurred during the study period. Room contamination was measured immediately before the application of the disinfectant (study day 0) and 24-hours later (day 1). Secondary outcomes included evaluation for clinically important pathogens (CIP), including methicillin-resistant staphylococcus aureus (MRSA), vancomycin-resistant Enterococcus (VRE) and carbapenem-resistant Enterobacteriaceae (CRE)

ELIGIBILITY:
Inclusion Criteria:

* Inpatient rooms housing adult patients on contact precautions

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Total room contamination | Day 1
  Total contamination, in colony-forming units (CFUs) on environmental surfaces on study day 1

SECONDARY OUTCOMES:
Clinically important pathogens (CIPs) in samples | Day 0
  Proportion of samples positive for individual CIP
Clinically important pathogens (CIPs) in samples | Day 1
  Proportion of samples positive for individual CIP
Baseline contamination (CFUs and CIPs) of sample areas | Day 0
  Similarity of baseline contamination measured in CFUs and proportion of samples positive for CIPs between sample area sides on study day 0 before application of the intervention
Compliance of routine disinfection | Day 1
  Proportion of sample areas with removed ultraviolet glowing gel on study day 1

CONTACTS AND LOCATIONS:
Overall Officials: Nick Turner, MD, Principal Investigator — Duke School of Medicine
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be reported in aggregate.

REFERENCES:
- [Derived] Warren BG, Barrett A, Graves A, King C, Turner NA, Anderson DJ. An Enhanced Strategy for Daily Disinfection in Acute Care Hospital Rooms: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2242131. doi: 10.1001/jamanetworkopen.2022.42131. PMID 36378308